CLINICAL TRIAL: NCT00399126
Title: A Phase 1 Trial of the Combination of Perifosine and Paclitaxel Given Either Weekly or Every 3 Weeks
Brief Title: Phase I Trial of Paclitaxel With Perifosine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 104
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2011-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — perifosine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Perifosine — Perifosine oral dose
Drug: Paclitaxel — Paclitaxel IV

SUMMARY:
This is a study of the drug perifosine given in combination with paclitaxel. Perifosine is an oral anti-cancer agent that has been used in more than 140 people. Paclitaxel is a standard chemotherapy agent used in many types of cancer. This study is designed to determine the highest dose of perifosine that can be administered to people every day while they are receiving paclitaxel in one of two regimens, without severe or prolonged nausea, vomiting and diarrhea. This study starts with patients taking 50 mg/day and goes up to 150 mg/day.

DETAILED DESCRIPTION:
This is a phase 1, open-label trial of perifosine and paclitaxel administered either weekly or every 3 weeks in patients with malignancies for whom single agent paclitaxel is a reasonable treatment option. All patients will receive paclitaxel either at a dose of 80 mg/m2 on days 1, 8 and 15 of a 28-day cycle (Arm A) or at 175 mg/m2 administered on day 8 of a 21 day cycle (Arm B). Patients on both arm A and arm B will receive premedication with diphenhydramine 50 mg IV 30 minutes prior to treatment; ranitidine 50 mg IV 30 minutes prior to treatment and dexamethasone 20 mg IV at 30 minutes prior to treatment. The 1st cohort of patients on Arm A will receive perifosine orally at a dose of 50 mg per day for the first 21 days of the 28-day cycle and on Arm B will receive perifosine orally at a dose of 50 mg per day for the first 14 days of the 21-day cycle. On each arm, the perifosine dose will be escalated in subsequent groups to 50 mg bid and then 50 mg tid as tolerated. (See below) Alternating cohorts of 3 patients will be entered first to Arm A and then to Arm B. The perifosine dose escalation for Arm A and Arm B will be performed separately according to the following algorithm. For each arm, a maximum tolerated dose (MTD) will be defined as a dose that can be given without grade 3/4 non-hematologic toxicity in more than 1/3 patients. If 2/3 patients in any cohort encounter a grade 3/4 non-hematologic toxicity, an additional 3 patients will be added. If the dose is intolerable for >3/6 patients then the previous dose level will be declared the MTD for that arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of cancer for which treatment with single agent paclitaxel would be an appropriate treatment option.
* At least 18 years of age.
* Patients can have received no more than two prior chemotherapy regimens for metastatic disease. Patients may be currently receiving paclitaxel using one of the schedules in the protocol, as long as the treating investigator has reasonable expectation that the patient will continue to receive paclitaxel for 2 or more additional cycles. The current regimen does not count towards the 2 regimens as long as the patient is not progressing on therapy.
* Patients must have a life expectancy of more than 3 months.
* Patients must have a performance status of 0 to 2 according to the ECOG criteria.
* Patients must have normal organ and marrow function as defined below: leukocytes >= 4,000/microL, absolute neutrophil count >= 1,500/microL, platelets >= 100,000/microL, HCT > 28%, total bilirubin < 2 x upper limit of normal, AST (SGOT)/ALT (SGPT) <= 2.5 X institutional upper limit of normal, creatinine <= 2.5 mg/dl transaminase < 2.5 times institution's upper normal limits
* Patients must have recovered from acute toxicity related to prior therapy, excluding alopecia, including surgery or radiotherapy.
* Patients must be able to ingest oral medications.
* Female patients who are pregnant or lactating are ineligible. All females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment. Men and women of childbearing potential must agree to employ adequate contraception to prevent pregnancy while on therapy and for four weeks after the completion of treatment.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents or devices.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Assoc. class II-IV congestive heart failure.
* Patients with a history of hypersensitivity reaction to products containing a Chremophor EL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-11; Primary Completion 2009-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
GI Toxicities | 3 months

SECONDARY OUTCOMES:
Other toxicities | 3 months
Disease progression | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- AOI Pharmaceuticals Investigative Site, Johnson City, Tennessee, United States

REFERENCES:
- [Result] 1) Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 24, No 18S (June 20 Supplement), 2006: 13134 2) Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 24, No 18S (June 20 Supplement), 2006: 13117